CLINICAL TRIAL: NCT00836862
Title: Arteriovenous Fistula Tissue Bank for Pre- and Post-Fistula Placement Specimens
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0482-08-EP
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Kidney Failure, Chronic
Keywords: Hemodialysis; Vascular access; Arteriovenous fistula
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Whole Blood, Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arteriovenous Fistula: A tissue bank will be created to collect serum, whole blood, and vein specimens obtained from participants undergoing Arteriovenous Fistula (AVF) placement and revision. The planned specimen harvests will allow for both pre- and post-AVF placement specimens from both maturing and failing AVF.
  Interventions: Other: Biologic specimens

INTERVENTIONS:
Other: Biologic specimens — Banking of serum, DNA and tissue

SUMMARY:
This project will bank sera, DNA and vascular specimens from patients undergoing arteriovenous fistula creation and revision.

DETAILED DESCRIPTION:
Hemodialysis patients utilizing an arteriovenous fistula (AVF) for hemodialysis access are 10 times less likely to develop bacteremia than those patients utilizing a hemodialysis catheter. Because of this, a great focus has been on placing AVF in all patients undergoing hemodialysis. While AVF are relatively simple to place from a surgical standpoint, 30-60% of AVF will not mature adequately to be used for hemodialysis. In order to be utilized for hemodialysis, the blood flow in the vein used to create the AVF will need to increase by over 100 fold. In order to do so, the vein will need to dilate by more than 150%. AVF which fail to mature do not dilate, and the major histologic finding in these AVF has been neointimal hyperplasia. The factors (both circulating and tissue) which contribute to AVF maturation or failure are poorly understood, and investigations in this area are limited. Current studies in the literature have either described pre-AVF vein characteristics, or have looked at serum or tissue specimens following AVF failure. To date, no studies have looked at specimens from patients both before and after fistula placement, or described factors associated with fistula maturation. This project will bank sera, DNA and vascular specimens from patients undergoing arteriovenous fistula creation and revision.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years of age or greater
* Arteriovenous fistula placement for hemodialysis access scheduled within 30 days

Exclusion Criteria:

* Incompetent to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be eligible if they are 19 years of age or greater and have placement of an arteriovenous fistula planned witin 30 days.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2012-11-10 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Troy J Plumb, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States